CLINICAL TRIAL: NCT01290263
Title: Phase I/II Study of Amgen 386 With and Without Bevacizumab for Recurrent Glioblastoma
Brief Title: Amgen 386 for Recurrent Glioblastoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, David Reardon, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-185
Record Dates: First submitted 2011-01-09; First posted 2011-02-04 (Estimated); Results first posted 2017-05-25 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Glioblastoma Multiforme
Keywords: Glioblastoma; GBM; Brain Tumor; Glioma
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms; Glioma | interventions — trebananib; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Amgen 386 (Experimental): Cohort A will assess recurrent Glioblastoma Multiforme (GBM) patients who receive AMG 386 monotherapy at 30mg/kg every week. As of August 1, 2013, Cohort A was closed to new accrual following early interim analysis of first 10 participants enrolled on study. None of these patients had achieved stable disease or response at their initial evaluation after 1-2 months of study therapy. Therefore, study investigators and sponsor agreed that the level of single-agent anti-tumor activity associated with AMG386 for recurrent glioblastoma patients is most likely insufficient to satisfy the stopping rule for low efficacy outlined in Section 14.5 for Cohort A.
  Interventions: Drug: Amgen 386
- Amgen 386 and Bevacizumab (Experimental): Cohort B will assess recurrent Glioblastoma Multiforme(GBM) patients who receive AMG 386 plus bevacizumab. Because the maximum tolerated dose of this combination therapy has not yet been established, a 3x3 Phase I study was used to determine the maximum tolerated dose. As of June 6, 2014, the MTD was determined to be AMG386 30 mg/kg administered intravenously every week(dose level +1) in combination with bevacizumab at 10mg/kg administered intravenously every other week. As of July 25, 2014 the Cohort B, Phase II portion of the study was opened to accrual.
  Interventions: Drug: Amgen 386; Drug: Bevacizumab

INTERVENTIONS:
Drug: Amgen 386 — For Cohort A, AMG 386 will be administered intravenously at 30 mg/kg every week.
  For Cohort B Phase I, AMG 386 will be administered intravenously at beginning at starting dose level of 15 mg/kg every week.
  For Cohort B Phase II, AMG 386 will be administered intravenously at the maximum tolerated dose determined in the Phase I portion of the study every week.
  Other Names: Trebananib
Drug: Bevacizumab — The dose of bevacizumab will be 10 mg/kg and will be administered intravenously every other week.
  Other Names: Avastin
  Arms: Amgen 386 and Bevacizumab

SUMMARY:
Primary Objectives

Cohort A -- monotherapy:

To determine the efficacy of AMG 386 in participants with recurrent glioblastoma (GBM) as measured by 6-month progression-free survival (PFS6)

Cohort B - combination therapy:

Phase I To determine the maximum tolerated dose of AMG 386 in combination with bevacizumab given at 10mg/kg every 2 weeks in participants with recurrent glioblastoma.

Phase II To determine the efficacy of AMG 386 plus bevacizumab in participants with recurrent glioblastoma (GBM) as measured by 6-month progression-free survival (PFS6).

Secondary Objectives:

To evaluate radiographic response in both cohort populations. To evaluate overall survival in both cohort populations. To assess time-to-progression in both cohort populations. To investigate the safety profile in both cohort populations.

Exploratory Objectives:

To evaluate expression of factors associated with tumor angiogenesis using a multiples cytokine assay among participants undergoing therapy with AMG 386 with response to therapy and development of resistance.

This is an open-label Phase I/II study of AMG 386 monotherapy and AMG 386 in combination with bevacizumab. Two cohorts will accrue and will be assessed sequentially. Each cohort will enroll participants with recurrent GBM. Cohort A will assess recurrent GBM participants who receive AMG 386 monotherapy at 30 g/kg every week. (Cohort A initially accrued at a dose of 15mg/kg, but this was increased to 30 mg/kg every week following an amendment). Cohort B will assess recurrent GBM participants who receive weekly AMG 386 plus bi-weekly bevacizumab (10mg/kg). Cohort B will start with a Phase I component to determine the MTD of AMG 386 that is safe when used in combination with bevacizumab. AMG 386 is administered intravenously, and, when used in combination with intravenous bevacizumab, will be administered first.

Patients will be required to come to the clinic weekly for study drug administration.

For study purposes, a cycle of therapy will be 4 weeks. Treatment will continue until either evidence of progressive disease, unacceptable toxicity, non-compliance with study follow-up, or withdrawal of consent.

The estimated rate of accrual is 60 participants per year. The estimated date of accrual completion is 1.5 years from study initiation. The estimated date of study completion will be approximately 12 months from enrollment of the last study participant.

ELIGIBILITY:
Inclusion Criteria

* Signed informed consent approved by the Institutional Review Board prior to participant entry
* Age ≥ 18 years.
* Karnofsky ≥ 70%
* Participant must be able and willing to comply with study and/or follow-up procedures Participants must have histologically confirmed diagnosis of GBM patients with either grade III or IV malignant glioma are eligible to the Phase I portion of the study) and radiographic evidence of recurrence or disease progression (defined as either a greater than 25% increase in the largest bidimensional product of enhancement, a new enhancing lesion, or significant increase in T2 FLAIR) following prior therapy (i.e. chemotherapy, XRT, other investigational therapies).
* No more than 2 prior episodes of progressive disease (patients with more than 2 prior episodes of progressive disease are eligible for the Cohort B, Phase I portion of this study)
* An interval of at least 4 weeks (to start of study agent) between prior surgical resection or one week from stereotactic biopsy
* An interval of at least 12 weeks (to start of study agent) from the end of prior radiotherapy unless there is a new area of enhancement consistent with recurrent tumor outside of the radiation field, or there is histological confirmation of unequivocal tumor progression
* From the projected start of scheduled study treatment, the following time periods must have relapsed: 4 weeks (or 5 half lives, whichever is shorter) from any investigational agent, 4 weeks (or 5 half lives, whichever is shorter) from cytotoxic therapy (except 23 days for temozolomide and 6 weeks from nitrosoureas), 6 weeks from antibodies (or 5 half lives, whichever is shorter), or 4 weeks (or 5 half lives, whichever is shorter) from other anti-tumor therapies.
* Participants must have recovered to a grade 0 or 1 from the toxic effects of prior therapy (with the exception of lymphopenia, which is common after therapy with temozolomide, and alopecia).
* No evidence of hemorrhage on the baseline MRI or CT scan other than those that are ≤ grade 1 and either post-operative or stable on at least two consecutive scans. Clinical Labs - performed within 14 days prior to enrollment
* Hematocrit ≥ 29%, ANC ≥ 1,000 cells/μl, platelets ≥ 100,000 cells/μl ;
* Serum creatinine ≤ 1.5 mg/dl, serum SGOT and bilirubin ≤ 1.5 times upper limit of normal;
* PTT or aPTT ≤ 1.5 times upper limit of normal and INR ≤ 1.5
* Calculated creatinine clearance ≥ 40 mL/min according to the Cockcroft-Gault formula OR per 24 hour urine collection
* Urinary protein quantitative value of < 30 mg/dL in urinalysis or <1+ on dipstick, unless quantitative protein is < 1000 mg in a 24 hour urine sample;
* Participants of child-bearing potential who have not undergone a bilateral salpingo-oophorectomy and are sexually active must consent to use an accepted and highly effective non-hormonal method of contraception (i.e. double barrier method [e.g., condom plus diaphragm]) from signing the informed consent through 6 months after last dose of study drug.

Exclusion Criteria:

* Prior anti-angiogenic therapy targeting VEGF or VEGF receptor including prior bevacizumab.
* Prior AMG 386 therapy or other molecules that inhibit the angiopoietins or Tie2 receptor.
* Co-medication that may interfere with study results; e.g. immunosuppressive agents other than corticosteroids.
* Active infection requiring intravenous antibiotics
* Current or within 30 days prior to enrollment treatment with immune modulators such as systemic cyclosporine and tacrolimus.
* Current us of warfarin sodium or any other Coumadin-derivative anticoagulant. Participant must be off Coumadin-derivative anticoagulants for at least seven days prior to starting study drug. ow molecular weight heparin is allowed.
* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study other than supportive care or epidemiologic studies.
* Herbal preparations/medications are not allowed throughout the study. These herbal medications include, but are not limited to: St. John's wort, Kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, ginseng. Participants should stop using any herbal medications 7 days prior to first dose of study drug.
* History of clinically significant bleeding within 6 months of enrollment
* History of allergic reactions to bacterially produced proteins
* Known hypersensitivity to any component of bevacizumab (cohort B only)
* Known sensitivity to any of the products to be administered during dosing
* History of venous or arterial thromboembolism within 12 months prior to enrollment.
* Severe hepatic insufficiency (ongoing grade 3 or greater hepatic adverse events) or known active chronic hepatitis.
* Inadequately controlled hypertension (defined as systolic blood pressure >140 and/or diastolic blood pressure > 90 mmHg). The use of anti-hypertensive medications to control hypertension is permitted.
* Any prior history of hypertensive crisis or hypertensive encephalopathy
* Clinically significant cardiovascular disease within 12 months prior to enrollment, including myocardial infarction, unstable angina, grade 2 or greater peripheral vascular disease, cerebrovascular accident, transient ischemic attack, congestive heart failure, or arrhythmias not controlled by outpatient medication, percutaneous transluminal coronary angioplasty/stent.
* Evidence of bleeding diathesis or coagulopathy
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study enrollment or anticipation of need for major surgical procedure during the course of the study
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to study enrollment.
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study enrollment.
* Serious, non-healing wound, ulcer (including gastrointestinal), or bone fracture.
* Any condition which in the investigator's opinion makes the subject unsuitable for study participation.
* Pregnant (positive pregnancy test) or lactating. Refusal or inability to use highly effective means of contraception (men and women) in participants of child-bearing potential.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2010-12; Primary Completion 2015-07 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Reardon, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (6):
- United States (6):
  - University of California Los Angeles, Los Angeles, California
  - Massachusetts General Hosptial, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts, Worcester, Worcester, Massachusetts
  - New York - Presbyterian/Columbia University Medical Center, New York, New York
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: As of August 1, 2013, Cohort A was closed to new accrual following early interim analysis of first 10 participants enrolled on study showed insufficient efficacy per design.
Groups:
- Cohort A: AMG 386 30 mg/kg: Cohort A participants received AMG 386 intravenously (IV) at 30 mg/kg on days 1, 8, 15 and 22 of each 28 day cycle. Participants were treated until disease progression or unacceptable toxicity.
- Cohort B Phase I Dose Level 0: AMG 386 15 mg/kg + Bevacizumab: Cohort B Phase I Dose Level 0 participants received bevacizumab 10 mg/kg intravenously (IV) on days 1 and 15 of each 28 day cycle and the original starting dose AMG 386 of 15 mg/kg intravenously (IV) on days 1, 8, 15 and 22. Participants were treated until disease progression or unacceptable toxicity.
- Cohort B Phase I Dose Level +1: AMG 386 30 mg/kg + Bevacizumab: Cohort B Phase I Dose Level +1 participants received bevacizumab 10 mg/kg intravenously (IV) on days 1 and 15 of each 28 day cycle and AMG 386 of 15 mg/kg intravenously (IV) on days 1, 8, 15 and 22. Participants were treated until disease progression or unacceptable toxicity.
  As of June 2014, the maximum tolerated dose (MTD) of bevacizumab + AMG 386 was determined to be dose level +1, AMG 386 30 mg + kg.
- Cohort B Phase II: AMG 386 30 mg/kg + Bevacizumab: Participants received bevacizumab 10 mg/kg intravenously (IV) on days 1 and 15 of each 28 day cycle and the maximum tolerated AMG 386 dose established in the Phase I Cohort B study, AMG 386 of 30 mg/kg intravenously (IV) on days 1, 8, 15 and 22. Participants were treated until disease progression or unacceptable toxicity.
- All Cohort B Participants: AMG 386 + Bevacizumab: Phase I & II Cohort B participants received bevacizumab 10 mg/kg intravenously (IV) on days 1 and 15 of each 28 day cycle and the assigned AMG 386 dose of 15 mg/kg or 30 mg/kg intravenously (IV) on days 1, 8, 15 and 22. Participants were treated until disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Cohort A: AMG 386 30 mg/kg | Cohort B Phase I Dose Level 0: AMG 386 15 mg/kg + Bevacizumab | Cohort B Phase I Dose Level +1: AMG 386 30 mg/kg + Bevacizumab | Cohort B Phase II: AMG 386 30 mg/kg + Bevacizumab | All Cohort B Participants: AMG 386 + Bevacizumab
Started | 11 | 3 | 7 | 27 | 37
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 11 | 3 | 7 | 27 | 37
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 1
Not completed — Lack of Efficacy | 8 | 2 | 7 | 24 | 33
Not completed — Withdrawal by Subject | 3 | 1 | 0 | 1 | 2
Not completed — Participant Non-Compliance | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Cohort B: AMG 386 + Bevacizumab: All Phase I & II Cohort B participants received bevacizumab 10 mg/kg intravenously (IV) on days 1 and 15 of each 28 day cycle and the assigned AMG 386 dose of 15 mg/kg or 30 mg/kg intravenously (IV) on days 1, 8, 15 and 22. Participants were treated until disease progression or unacceptable toxicity.
- Cohort A: AMG 386 30 mg/kg: All cohort A participants received AMG 386 intravenously (IV) at 30 mg/kg on days 1, 8, 15 and 22 of each 28 day cycle. Participants were treated until disease progression or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | Cohort B: AMG 386 + Bevacizumab | Cohort A: AMG 386 30 mg/kg | Total
Number analyzed (Participants) | 37 | 11 | 48
Age, Continuous [Median (Full Range); unit: years] | 63 [37 to 86] | 62 [29 to 78] | 62 [29 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 5 | 16
  Male | 26 | 6 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 35 | 10 | 45
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 35 | 10 | 45
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 1 | 0 | 1
Number of Prior Relapses [Number; unit: participants]
  1 | 23 | 8 | 31
  2 | 14 | 2 | 16
  3 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: 6-Month Progression-Free Survival (PFS6) [Cohort A and Cohort B]
Description: PFS6 is the proportion of patients remaining alive and progression-free at 6-months from study entry. Progressive disease was established based on Response Assessment in Neuro-Oncology (RANO) criteria (Wen et al JCO 2010). RANO criteria has 5 potential categories: Complete Response (CR), Partial Response (PR), Stable Disease (SD), Progressive disease (PD) and Unknown status. CR: disappearance of all enhancing lesions, stable or improved non-enhancing lesions, and stable or improved clinically. PR: >= 50% decrease in sum of perpendicular diameters of all measurable enhancing lesions, no progression of non-measurable disease, stable or improved non- enhancing lesions, and stable or improved clinically. PD: > 25% increase in sum of perpendicular diameters of all measurable enhancing lesions, significant increase of non-enhancing lesions, any new lesions, clear clinical deterioration, failure to return for evaluation due to death or deteriorating condition. SD: d
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- All Cohort B Participants: AMG 386 + Bevacizumab: All Phase I & II Cohort B participants received bevacizumab 10 mg/kg intravenously (IV) on days 1 and 15 of each 28 day cycle and the assigned AMG 386 dose of 15 mg/kg or 30 mg/kg intravenously (IV) on days 1, 8, 15 and 22. Participants were treated until disease progression or unacceptable toxicity.
Arm/Group | All Cohort B Participants: AMG 386 + Bevacizumab | Cohort A: AMG 386 30 mg/kg
Number analyzed (Participants) | 37 | 11
proportion of participants | 0.243 [0.12 to 0.38] | 0 [0 to 0]

2. Primary Outcome: AMG 386 Maximum Tolerated Dose (MTD) [Cohort B Phase I]
Description: The MTD of weekly AMG 386 intravenously (IV) in combination with bevacizumab 10 mg/kg intravenously (IV) on days 1 and 15 of each 28 day cycle is determined by the number of participants who experience a dose limiting toxicity (DLT). See subsequent primary outcome measure for the DLT definition. The MTD is defined as the highest dose at which fewer than one-third of patients experience a DLT. If no DLTs are observed, the MTD is not reached but the highest dose received may be the Recommended Phase II Dose (RP2D).
Time Frame: Participants were assessed weekly while on study; the observation period for MTD evaluation was the first 28 days of study treatment.
Population: All phase I Cohort B participants who received at least one dose of the study drug were evaluable for MTD. A participant was replaceable if they are taken off of study treatment due to progressive disease or withdrawal from study during before they completed the 28 day DLT period.
Measure: Number; unit: mg/kg intravenously on days 1 and 15
Groups:
- Cohort B Phase I Dose Level +1: AMG 386 30 mg/kg + Bevacizumab: Cohort B Phase I Dose Level +1 participants received bevacizumab 10 mg/kg intravenously (IV) on days 1 and 15 of each 28 day cycle and AMG 386 of 15 mg/kg intravenously (IV) on days 1, 8, 15 and 22. Participants were treated until disease progression or unacceptable toxicity.
  As of June 2014, the maximum tolerated dose (MTD) of bevacizumab + AMG 386 was determined to be dose level +1, AMG 386 30 mg/kg.
Arm/Group | Cohort B Phase I Dose Level 0: AMG 386 15 mg/kg + Bevacizumab | Cohort B Phase I Dose Level +1: AMG 386 30 mg/kg + Bevacizumab
Number analyzed (Participants) | 3 | 7
mg/kg intravenously on days 1 and 15 | 30 | 30

3. Secondary Outcome: Best Radiographic Response [Cohort A and Cohort B]
Description: Radiographic response was established based on Response Assessment in Neuro-Oncology (RANO) criteria (Wen et al JCO 2010) with 5 potential categories: Complete Response (CR), Partial Response (PR), Stable Disease (SD), Progressive disease (PD) and Unknown status. CR: disappearance of all enhancing lesions, stable or improved non-enhancing lesions, and stable or improved clinically. PR: >= 50% decrease in sum of perpendicular diameters of all measurable enhancing lesions, no progression of non-measurable disease, stable or improved non- enhancing lesions, and stable or improved clinically. PD: > 25% increase in sum of perpendicular diameters of all measurable enhancing lesions, significant increase of non-enhancing lesions, any new lesions, clear clinical deterioration, failure to return for evaluation due to death or deteriorating condition. SD: does not qualify for CR, PR or PD, stable non-enhancing lesions, and stable clinically.
Time Frame: Disease was assessed radiographically for response every 8 weeks.
Population: All participants who received at least one dose of the study drug were evaluable for response.
Measure: Number; unit: participants
Arm/Group | All Cohort B Participants: AMG 386 + Bevacizumab | Cohort A: AMG 386 30 mg/kg
Number analyzed (Participants) | 37 | 11
participants
  Complete Response | 0 | 0
  Partial Response | 4 | 0
  Stable Disease | 20 | 1
  Progressive Disease | 10 | 8
  Unknown | 3 | 2

4. Secondary Outcome: Overall Survival (OS) [Cohort A and Cohort B]
Description: OS based on Kaplan-Meier is defined as the time from study entry to death or date last known alive.
Time Frame: Participants were followed long-term for survival every 3 to 4 months from the end of treatment until death or lost to follow-up. On Cohort A and B participants were followed up to 554 days and 442 days.
Population: All participants who received at least one dose of the study drug were followed for OS.
Measure: Median (Full Range); unit: days
Arm/Group | All Cohort B Participants: AMG 386 + Bevacizumab | Cohort A: AMG 386 30 mg/kg
Number analyzed (Participants) | 37 | 11
days | 285 [225 to 442] | 341 [138 to 554]

5. Secondary Outcome: Progression-Free Survival (PFS) [Cohort A and Cohort B]
Description: PFS based on Kaplan-Meier is defined as the time from study entry to the earliest documentation of disease progression or death. Progressive disease was established based on Response Assessment in Neuro-Oncology (RANO) criteria (Wen et al JCO 2010).
Time Frame: Disease was assessed radiographically to document clinical progression every cycle on treatment and post-treatment every 8 weeks. On Cohort A and B participants were followed for progression up to 36 days and 166 days.
Population: All participants who received at least one dose of the study drug were evaluable for PFS.
Measure: Median (Full Range); unit: days
Arm/Group | All Cohort B Participants: AMG 386 + Bevacizumab | Cohort A: AMG 386 30 mg/kg
Number analyzed (Participants) | 37 | 11
days | 108 [56 to 166] | 21 [5 to 36]

6. Primary Outcome: AMG 386 Dose Limiting Toxicity (DLT) [Cohort B Phase I]
Description: A DLT is defined as an adverse event that (a) is related to the AMG 386 and/or bevacizumab with an attribution of possible, probable, or definite, and (b) occurs during and/or begins during the first 28 days of the study treatment, and (c) meets any of the following criteria: >= grade 3 thrombocytopenia; grade 4 neutropenia lasting > 7 days; grade 4 anemia lasting > 7 days despite transfusion or growth factors; febrile neutropenia if ANC<0.5x10^9/L; clinically significant grade 3 non-hematologic toxicity despite maximal medical therapy lasting > 7 days, with the exception of grade 3 proteinuria which was considered a DLT if lasting > 14 days; grade 3 non-hematologic toxicity resulting in study drug discontinuation; grade 4 non-hematologic toxicity; >= grade 1 new CNS hemorrhage; >= grade 2 non-CNS hemorrhage.
Time Frame: Participants were assessed weekly while on study; the observation period for DLT evaluation was the first 28 days of study treatment.
Population: All phase I Cohort B participants who completed 28 days on study treatment were evaluable. A participant was replaceable if they are taken off of study treatment due to progressive disease or withdrawal from study during before they completed the 28 day DLT period.
Measure: Number; unit: participants
Arm/Group | Cohort B Phase I Dose Level 0: AMG 386 15 mg/kg + Bevacizumab | Cohort B Phase I Dose Level +1: AMG 386 30 mg/kg + Bevacizumab
Number analyzed (Participants) | 3 | 7
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Assessed each treatment cycle (1 cycle = 28 days) from time of first dose and up to day 30 post-treatment. Treatment duration in cycles was a median (range) of 1 (1-2) Cohort A and 4 (1-20) Cohort B.
Description: Maximum grade toxicity by type was first calculated. Serious AEs were defined as events with AMG386 and/or bevacizumab treatment-attribution of at least possibly and causing a hospitalization, deemed serious by the treating investigator or grade 5 events per CTCAE v4. Other AEs were defined as events with AMG386 and/or bevacizumab treatment-attribution of at least possibly and not requiring a hospitalization or deemed non-serious by treating investigator.
Arm/Group | Cohort B: AMG 386 + Bevacizumab | Cohort A: AMG 386 30 mg/kg
Serious Adverse Events (participants affected / at risk) | 5/37 | 0/11
Other Adverse Events (participants affected / at risk) | 30/37 | 8/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort B: AMG 386 + Bevacizumab (N=37) | Cohort A: AMG 386 30 mg/kg (N=11)
Platelet count decreased (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Grade 4 Platelet count decreased
Edema Limbs (General disorders) | 1 (1) | 0 (0) — Grade 3 Edema Limbs
Fatigue (General disorders) | 1 (1) | 0 (0) — Grade 3 Fatigue
Fatigue (General disorders) | 1 (1) | 0 (0) — Grade 2 Fatigue
Neutrophil Count Decreased (Investigations) | 1 (1) | 0 (0) — Grade 4 Neutrophil Count Decreased
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort B: AMG 386 + Bevacizumab (N=37) | Cohort A: AMG 386 30 mg/kg (N=11)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) — Grade 2 Anemia
Atrial Flutter (Cardiac disorders) | 1 (1) | 0 (0) — Grade 2 Atrial Flutter
Pericardial Effusion (Cardiac disorders) | 1 (1) | 0 (0) — Grade 2 Pericardial Effusion
Blurred Vision (Eye disorders) | 0 (0) | 1 (1) — Grade 1 Blurred Vision
Blurred Vision (Eye disorders) | 1 (1) | 0 (0) — Grade 2 Blurred Vision
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 1 (1) — Grade 1 Abdominal Pain
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) — Grade 2 Abdominal Pain
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) — Grade 1 Constipation
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) — Grade 2 Constipation
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) — Grade 1 Diarrhea
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) — Grade 2 Diarrhea
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) — Grade 1 Dry Mouth
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) — Grade 1 Hemorrhoids
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (2) — Grade 1 Nausea
Stomach Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) — Grade 1 Stomach Pain
Edema Face (General disorders) | 1 (1) | 0 (0) — Grade 1 Edema Face
Edema Limbs (General disorders) | 3 (3) | 1 (1) — Grade 1 Edema Limbs
Edema Limbs (General disorders) | 2 (2) | 0 (0) — Grade 2 Edema Limbs
Fatigue (General disorders) | 3 (3) | 0 (0) — Grade 1 Fatigue
Fatigue (General disorders) | 3 (3) | 2 (2) — Grade 2 Fatigue
Infusion Related Reaction (General disorders) | 1 (1) | 0 (0) — Grade 2 Infusion Related Reaction
Infusion Site Reaction (General disorders) | 1 (1) | 0 (0) — Grade 1 Infusion Site Reaction
Localized Edema (General disorders) | 1 (1) | 0 (0) — Grade 2 Localized Edema
Gait Disturbance (General disorders) | 0 (0) | 1 (1) — Grade 1 Gait Disturbance
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Grade 1 Bruising
Vascular Access Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Grade 2 Vascular Access Complication
Alanine Aminotransferase Increased (Investigations) | 2 (2) | 0 (0) — Grade 1 Alanine Aminotransferase Increased
Alkaline Phosphatase Increased (Investigations) | 1 (1) | 0 (0) — Grade 1 Alkaline Phosphatase Increased
Aspartate Aminotransferase Increased (Investigations) | 2 (2) | 0 (0) — Grade 1 Aspartate Aminotransferase Increased
Blood Bilirubin Increased (Investigations) | 1 (1) | 0 (0) — Grade 1 Blood Bilirubin Increased
Cardiac Troponin I Increased (Investigations) | 1 (1) | 0 (0) — Grade 3 Cardiac Troponin I Increased
Neutrophil Count Decreased (Investigations) | 1 (1) | 0 (0) — Grade 1 Neutrophil Count Decreased
Neutrophil Count Decreased (Investigations) | 1 (1) | 0 (0) — Grade 2 Neutrophil Count Decreased
Platelet Count Decreased (Investigations) | 4 (4) | 0 (0) — Grade 1 Platelet Count Decreased
Platelet Count Decreased (Investigations) | 1 (1) | 0 (0) — Grade 4 Platelet Count Decreased
White Blood Cell Decreased (Investigations) | 1 (1) | 0 (0) — Grade 1 White Blood Cell Decreased
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Grade 1 Anorexia
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) — Grade 1 Hyperglycemia
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) — Grade 1 Hypokalemia
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) — Grade 1 Hyponatremia
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Grade 3 Hypophosphatemia
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) — Grade 1 Arthralgia
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) — Grade 1 Generalized Muscle Weakness
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Grade 2 Muscle Weakness Lower Limb
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Grade 1 Myalgia
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) — Grade 1 Dizziness
Headache (Nervous system disorders) | 2 (2) | 1 (1) — Grade 1 Headache
Intracranial Hemorrhage (Nervous system disorders) | 1 (1) | 0 (0) — Grade 1 Intracranial Hemorrhage
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) — Grade 1 Presyncope
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) — Grade 1 Confusion
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) — Grade 1 Insomnia
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) — Grade 2 Insomnia
Hematuria (Renal and urinary disorders) | 3 (3) | 0 (0) — Grade 1 Hematuria
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) — Grade 1 Proteinuria
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) — Grade 2 Proteinuria
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) — Grade 1 Epistaxis
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (1) — Grade 1 Hoarseness
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) — Grade 1 Alopecia
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Grade 1 Rash Maculo-papular
Skin Ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Grade 1 Skin Ulceration
Hypertension (Vascular disorders) | 2 (2) | 0 (0) — Grade 1 Hypertension
Hypertension (Vascular disorders) | 10 (10) | 0 (0) — Grade 2 Hypertension
Hypertension (Vascular disorders) | 3 (3) | 0 (0) — Grade 3 Hypertension
Thromboembolic Event (Vascular disorders) | 2 (2) | 0 (0) — Grade 2 Thromboembolic Event
Thromboembolic Event (Vascular disorders) | 1 (1) | 0 (0) — Grade 3 Thromboembolic Event
Other - Conjunctival Hemorrhage (Eye disorders) | 1 (1) | 0 (0) — Grade 1 Other - Conjunctival Hemorrhage
Other - Indigestion/heartburn (Gastrointestinal disorders) | 0 (0) | 1 (1) — Grade 2 Other - Indigestion/heartburn
Other - Livedo Reticularis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Grade 1 Other - Livedo Reticularis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No